CLINICAL TRIAL: NCT01567748
Title: In-human Validation of a Technique for Measuring Central Aortic Hemodynamics With Peripheral Arterial Waveforms
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Barry Finegan, Principal Investigator, Clinical Professor, Department of Anesthesiology, University of Alberta
Other Study IDs: 00021889
Record Dates: First submitted 2012-02-14; First posted 2012-03-30 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Coronary Artery Disease
Keywords: CABG; Coronary Artery Bypass; Central Aortic Pressure; Peripheral Arterial Waveform
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hemodynamics Measured: The following additional research related procedures will be performed in patients recruited into the study: 1) a small cuff will be placed on one the finger of each subject to measure the pulse in the finger (Finapres); 2) a cannula will be placed in the femoral artery by the surgeon to measure femoral artery pressure; 3) for a period of two minutes immediately before and after the cardiopulmonary bypass a small cannula (the size of a pencil tip) will be inserted by the surgeon under direct vision into the aorta and 4) the information from each of these cannula will be recorded on a computer for later study.
  Interventions: Procedure: BP Measurements at aorta, radial and femoral locations

INTERVENTIONS:
Procedure: BP Measurements at aorta, radial and femoral locations — The following additional research related procedures will be performed in patients recruited into the study: 1) a small cuff will be placed on one the finger of each subject to measure the pulse in the finger (Finapres); 2) a cannula will be placed in the femoral artery by the surgeon to measure femoral artery pressure; 3) for a period of two minutes immediately before and after the cardiopulmonary bypass a small cannula (the size of a pencil tip) will be inserted by the surgeon under direct vision into the aorta and 4) the information from each of these cannula will be recorded on a computer for later study.

SUMMARY:
Central aortic blood pressure (BP) and flow are generally more informative about the health condition of the heart and the arterial system compared with BP measured in peripheral locations (e.g. arm or leg). However, their clinical impact has been limited due to the cost, risk and discomfort associated with their measurements. Peripheral BP is attractive because it can be measured relatively easily than central aortic BP. However, peripheral BP is not as useful as central aortic BP since the shape of its waveform is different from that of central aortic BP. The applicant recently developed two innovative methods, the "Individualized Transfer Functions (ITF)," which is able to estimate the central aortic BP waveform of a patient using the measurements of peripheral BP waveform(s). The methods were successfully validated using animal and simulated human subjects. The objective of the proposed research project is to examine the validity of these innovative methods in human subjects.

Cardiovascular disease accounts for 1/3 of all deaths and more than $22 billion healthcare-related cost in Canada every year. The proposed research project will make significant contribution in improving clinical care by the potential of ITF in detection and diagnostics of cardiovascular disease. In fact, the proposed research project is a key initial step towards our long-term research objective of non-invasive cardiovascular disease diagnostics. The success of the proposed research project will demonstrate that ITF can serve as a low-cost, non-invasive and convenient alternative for central aortic BP measurement, which can further be used for the development of detection and diagnostics methods for a number of cardiovascular diseases (e.g. aortic valve impairment and peripheral arterial disease) by virtue of the relevant health and disease conditions of central and peripheral arterial vessels that ITF can deliver.

DETAILED DESCRIPTION:
Central aortic blood pressure (BP) and flow are generally more informative about cardiac dynamics and global circulation compared with cardiovascular parameters measured in the periphery [1,2]. However, their clinical impact has been limited due to significant clinical risk and substantial cost associated with their measurements. Peripheral arterial BP's are easily obtained non-invasively, but they cannot serve as direct substitutes for central aortic BP due to the distortion of arterial BP waveform caused by pressure wave propagation and reflection. Recently, two innovative model-based methods, the "Individualized Transfer Functions (ITF)," have been developed by Dr. Hahn to estimate central aortic BP waveform using the measurements of peripheral BP waveform(s) [3-6]. These techniques have been validated in animal and simulated human subjects. The objective of the proposed research project is to 1) examine the feasibility and validity of these innovative methods in human subjects, and 2) compare the performance of these methods against direct peripheral BP and existing non-individualized (NITF) methods.

The proposed research project consists of two major parts: 1) collection of central aortic and peripheral BP data, and 2) evaluation of ITF methods using these data. BP data will be collected from the patients already undergoing procedures with cardiopulmonary bypass. Central aortic, radial and femoral BP waveforms will be simultaneously recorded. A non-invasive finger BP waveform will also be recorded. The pair of radial-femoral or finger-femoral BP recordings will be analyzed by the two-measurement ITF [3-5] to estimate individual-specific central aortic BP waveform. In addition, radial or finger BP recording will be analyzed by the single-measurement ITF [6] to estimate individual-specific central aortic BP waveform. The feasibility and validity of the methods in human subjects will be assessed by comparing the estimated central aortic BP waveforms with the measured central aortic BP waveforms. Its relative performance with respect to direct peripheral BP and existing NITF methods will be analyzed by comparing the difference between measured central aortic versus ITF-derived central aortic BP waveforms with those between measured central aortic versus direct peripheral and NITF-derived central aortic BP waveforms.

Cardiovascular disease accounts for 1/3 of all deaths and more than $22 billion healthcare-related cost in Canada every year [7]. The proposed research project will make significant contribution in improving clinical care through the use of ITF in detection and diagnostics of cardiovascular disease. In fact, the proposed research project is a key initial step towards our long-term research objective of non-invasive cardiovascular disease diagnostics. The success of the proposed research project will be a milestone to demonstrate that ITF can serve as minimally invasive and/or non-invasive approach whose individually estimated central aortic BP waveform and cardiovascular system model can be exploited for detection and diagnostics of a number of cardiovascular disease, e.g. aortic valve impairment and peripheral arterial disease, by virtue of diagnostically relevant health and disease conditions of central and peripheral arterial vessels that ITF can deliver.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18 through 80 years, inclusive
* Scheduled for coronary artery bypass surgery with CPB

Exclusion Criteria:

* Scheduled for heart surgery other than coronary artery bypass surgery
* Females of childbearing potential
* Emergency surgery
* BMI > 35

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is looking at those individuals undergoing Coronary Artery Bypass surgery requiring CPB, between the age of 18-80, with a BMI < 35.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Validate ITF Methodology | Intra Operatively
  We will collect the relevant circulatory (BP) data and apply these data to validate the Individualized Transfer Function (ITF) methodology

CONTACTS AND LOCATIONS:
Overall Officials: Barry A Finegan, MB, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital/Mazankowski Alberta Heart Institute, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Safar ME, Jankowski P. Central blood pressure and hypertension: role in cardiovascular risk assessment. Clin Sci (Lond). 2009 Feb;116(4):273-82. doi: 10.1042/CS20080072. PMID 19138169
- [Background] Papaioannou TG, Protogerou AD, Stamatelopoulos KS, Vavuranakis M, Stefanadis C. Non-invasive methods and techniques for central blood pressure estimation: procedures, validation, reproducibility and limitations. Curr Pharm Des. 2009;15(3):245-53. doi: 10.2174/138161209787354203. PMID 19149616
- [Background] J.O. Hahn et al., 2009, ASME Journal of Dynamic Systems, Measurement and Control 131: 051009
- [Background] J.O. Hahn et al., 2009, Control Engineering Practice 17: 1318-1328
- [Background] Hahn JO, Reisner AT, Asada HH. Estimation of pulse transit time using two diametric blood pressure waveform measurements. Med Eng Phys. 2010 Sep;32(7):753-9. doi: 10.1016/j.medengphy.2010.04.017. Epub 2010 May 26. PMID 20537933